CLINICAL TRIAL: NCT02529228
Title: Combined Effects of Meal Frequency and Protein Load on Cardiometabolic Risk Factors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore Institute of Food and Biotechnology Innovation (Other Government)
Responsible Party: Principal Investigator, Melvin Leow, Principal Investigator, Singapore Institute of Food and Biotechnology Innovation
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 2015/01504
Record Dates: First submitted 2015-08-17; First posted 2015-08-20 (Estimated); Last update posted 2015-08-20 (Estimated); Status verified 2015-08

CONDITIONS: Metabolic Disease; Cardiovascular Disease
MeSH Terms: conditions — Metabolic Diseases; Cardiovascular Diseases | interventions — Meals; Eating; RFC3 protein, Arabidopsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- CON-2 (Experimental): Consuming 2 Low Protein, High Carbohydrate Meals i.e. changing Meal Frequency and Protein Composition.
  Interventions: Other: Meal (Eating) Frequency; Other: Protein Composition
- CON-6 (Experimental): Dividing meal intake into 6 smaller Low Protein, High Carbohydrate Meals. i.e. changing Meal Frequency and Protein Composition.
  Interventions: Other: Meal (Eating) Frequency; Other: Protein Composition
- PRO-2 (Experimental): Consuming 2 High Protein, Low Carbohydrate Meals. i.e. changing Meal Frequency and Protein Composition.
  Interventions: Other: Meal (Eating) Frequency; Other: Protein Composition
- PRO-6 (Experimental): Dividing meal intake into 6 smaller High Protein, Low Carbohydrate Meals. i.e. changing Meal Frequency and Protein Composition.
  Interventions: Other: Meal (Eating) Frequency; Other: Protein Composition

INTERVENTIONS:
Other: Meal (Eating) Frequency — Dividing meal intake into 2 or 6 meals with equal energy content
Other: Protein Composition — Consuming meals with higher or lower protein.

SUMMARY:
This study examines the effect of meal frequency and meal composition on risk factors of cardiometabolic disease.

DETAILED DESCRIPTION:
Cardio-Metabolic Disease (CMD) is the leading cause of death globally & in Singapore. Large scale epidemiological evidence confirmed that elevated postprandial Glucose, Insulin, Triglycerides are major risk factors for CMD. Recent evidence suggests benefits from high protein diets but the health effects of eating smaller meals remain enigmatic. The aim of this study is to examine Meal frequency (2-large vs 6-smaller isocaloric meals), under High or Low Protein loads on acute postprandial health biomarkers . The investigators hypothesized that Higher Protein & Higher Meal Frequency would be beneficial for cardiometabolic health.

ELIGIBILITY:
Inclusion Criteria:

* Chinese Males
* Age: 21 - 50 years.
* Body mass stable within the last 2 months by self-report.
* Body mass index (BMI): < 30kg/m2.
* Normal fasting blood glucose level≤ 6.0 mmol/L
* Blood pressure ≤ 140/90 mmHg
* Not participating in any dietary interventions in the past 2-months.

Exclusion Criteria:

* Special dietary practice (e.g. Vegetarians, Atkins diet) or diets due to religious reasons during the study period (e.g. Fasting for Ramadan)
* Smoking.
* Excessive alcohol consumption: consuming alcohol on >4 days per week with ≥5 alcoholic drinks (males) and ≥4 alcoholic drinks (females) per time (National Health Survey, 2010).
* Metabolic Diseases (including thyroid dysfunction)
* Using Medication affecting carbohydrate and fat metabolism
* Allergy to any components of the provided meals (gluten, nuts, milk, dairy)

Ages: 21 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2014-12; Primary Completion 2015-05 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Venous Plasma Glucose | Postprandially 8.5 hours in response to the various diets
  Biochemical variable on a continuous scale.
Venous Plasma Insulin | Postprandially 8.5 hours in response to the various diets
  Biochemical variable on a continuous scale.
Venous Plasma Triglyceride | Postprandially 8.5 hours in response to the various diets
  Biochemical variable on a continuous scale.
Blood Pressure | Postprandially 8.5 hours in response to the various diets
  Systolic and Diastolic Pressure measured in mmHg
Interstitial Glucose | Postprandially 8.5 hours in response to the various diets
  Measured using a continuous glucose monitor.

SECONDARY OUTCOMES:
Urinary F2 Isoprostanes | Postprandially 8.5 hours in response to the various diets
  Biochemical variable on a continuous scale.
Subjective Appetite Ratings | Postprandially 8.5 hours in response to the various diets
  Measured on a 100mm Visual Analog Scale (VAS). 0mm=Not full at all, 100mm= Extremely full.

REFERENCES:
- [Derived] Mok A, Haldar S, Lee JC, Leow MK, Henry CJ. Postprandial changes in cardiometabolic disease risk in young Chinese men following isocaloric high or low protein diets, stratified by either high or low meal frequency - a randomized controlled crossover trial. Nutr J. 2016 Mar 15;15:27. doi: 10.1186/s12937-016-0141-5. PMID 26979583